CLINICAL TRIAL: NCT02777918
Title: Changing Habits and Lifestyles in Older Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bournemouth University (Other)
Collaborators: British Egg Industry Council (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BUREC12036
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-06

CONDITIONS: Eating Behaviour
Keywords: food intake
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): 6 recipes will be sent by post every 2 weeks for a 12 week period. Dietary recommendations will also be provided at the start of the intervention period to increase the relevance of the recipes.
  Interventions: Behavioral: Recipe provision
- Control (No Intervention): Dietary recommendations will be provided at the start of the study period, such that the intervention regards the recipes, not the recommendations

INTERVENTIONS:
Behavioral: Recipe provision — 6 recipes will be provided every 2 weeks by post for 12 weeks
  Arms: Intervention

SUMMARY:
This is an intervention study, aiming to increase protein intake, by increasing egg consumption in community dwelling older adults aged 55 years and over, by providing recipes to increase flavour and variety in egg dishes.

DETAILED DESCRIPTION:
Individuals will be randomized to either receive the intervention or to a control group, where the intervention group will receive 6 recipes every two weeks for a 12 week period, and at the start, after 12 weeks and after 6 months egg intake, protein intake, body protein status, and various functional measures of muscle function will be assessed in both intervention and control group.

ELIGIBILITY:
Inclusion Criteria:

Individuals can be considered for inclusion if they meet the following inclusion criteria:

* being over 55 years old
* living in the community
* being able to give consent
* not being allergic to eggs
* not suffering from known renal insufficiency, or having a pacemaker or defibrillator.
* not suffering from known hypercholesterolaemia, or known familial hypercholesterolaemia.
* not having undergone chemotherapy or radiotherapy in the last 6 months
* not suffering from any condition, or receiving medication or treatment that the participants feel affects their eating or sense of flavour.
* being able to perform the physical performance tests (e.g. walk, sit on a chair)
* being able to read and understand English

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Appleton, PhD, Principal Investigator — Bournemouth University

IPD SHARING:
Plan to Share IPD: No
Group data will be made available on publication of the study

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 53 | 47
Completed | 50 | 43
Not Completed | 3 | 4
Not completed — Medical reasons | 1 | 2
Not completed — Too busy / stressed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 53 | 47 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (8) | 70 (7) | 70 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 24 | 54
  Male | 23 | 23 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 53 | 47 | 100

OUTCOME MEASURES:

1. Primary Outcome: Egg Intake
Description: Egg intake at the end of the intervention period, assessed using an adapted Food Frequency Questionnaire (FFQ)
Time Frame: Change from baseline to 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: eggs
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 47
eggs | 5 (20) | 4 (20)

2. Primary Outcome: Adverse Events
Description: Self-declared adverse events over the intervention period, assessed by questionnaire
Time Frame: Change from baseline to 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: Adverse events
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 47
Adverse events | 0.1 (1.9) | 0.3 (1.3)

3. Secondary Outcome: Change in Dietary Protein Intake
Description: Change in dietary protein intake over the intervention and follow-up period, assessed using an adapted FFQ
Time Frame: Change from baseline to 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: g/day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 47
g/day | -3 (29) | 3 (35)

4. Secondary Outcome: Muscle Function
Description: Muscle function over the intervention and follow-up period, assessed using the Short Physical Performance Battery (Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. (1994) A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol 49:M85-M94). Higher scores denote better ability - range - 5.0 to +5.0.
Time Frame: Change from baseline to 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 47
scores on a scale | 0.6 (2.6) | -0.2 (2.1)

5. Secondary Outcome: Lean Body Mass
Description: Lean body mass over the intervention and follow-up period, assessed using bioimpedance
Time Frame: Change from baseline to 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 47
g | -0.1 (12.6) | -0.3 (12.8)

6. Secondary Outcome: Egg Intake
Description: Egg intake over the follow-up period, assessed using an adapted FFQ.
Time Frame: 6 months
Population: ITT
Measure: Mean (Standard Deviation); unit: eggs
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 47
eggs | 4 (22) | 1 (15)

7. Secondary Outcome: Number of Adverse Events Reported
Description: Self-declared adverse events over the follow-up period, assessed by questionnaire
Time Frame: 6 months
Population: ITT
Measure: Mean (Standard Deviation); unit: Number of adverse events reported
Arm/Group | Intervention | Control
Number analyzed (Participants) | 53 | 47
Number of adverse events reported | 0.3 (1.5) | 0.5 (1.7)

ADVERSE EVENTS:
Time Frame: 6 months
Description: self-report questionnaire assessing number of unusual experiences of nausea, digestive issues (e.g. constipation or diarrhoea), stomach aches/cramps, hunger, bloating/uncomfortable fullness, thirst, headaches, fatigue/tiredness, restlessness, dizziness, or skin rashes.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/47
Other Adverse Events (participants affected / at risk) | 53/53 | 47/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=53) | Control (N=47)
Questionnaire self-report (General disorders) | 53 (53) | 47 (47) — Any unspecified general physical disorder

LIMITATIONS AND CAVEATS:
Anticipated, but small sample. Should be treated as a pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/18/NCT02777918/Prot_SAP_000.pdf